CLINICAL TRIAL: NCT02075385
Title: Randomized Phase II Trial: Swallowing Speech Pathology Intervention During Radiochemotherapy on Patients With Head and Neck Cancer
Brief Title: Swallowing Intervention During Radiochemotherapy on Head and Neck Cancer
Acronym: Swallowing-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 589/2012
Record Dates: First submitted 2014-01-23; First posted 2014-03-03 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2015-10

CONDITIONS: Head Neck Cancer; Swallowing Disorders
Keywords: Dysphagia; speech language therapy; quality of life; induction chemotherapy; concurrent chemoradiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders; Communication Disorders | interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Speech pathology therapy (Experimental): Pre, during and pos-treatment swallowing exercises.
  Interventions: Procedure: pre, during and pos-treatment swallowing exercises
- Control group (No Intervention): These patients will not receive speech pathology therapy.

INTERVENTIONS:
Procedure: pre, during and pos-treatment swallowing exercises — Speech pathology therapy
  Other Names: swallowing pathology therapy
  Arms: Speech pathology therapy

SUMMARY:
General Objective: To evaluate the swallowing results of speech pathologist rehabilitation of advanced oropharynges, larynx and hypopharynx cancer patients during neoadjuvant chemotherapy and radiotherapy concomitant to chemotherapy.

Methods and Casuistic: Randomized clinical trial phase II. 80 patients with advanced oropharynges, larynx and hypopharynx cancer diagnoses from Barretos Cancer Hospital, which had the proposal of neoadjuvant chemotherapy followed by radiotherapy combined with chemotherapy. Patients are randomized on two groups: control group and speech pathology therapy group

DETAILED DESCRIPTION:
To evaluate and compare the swallowing and life quality swallowing on a group undergoing to speech pathology therapy (intervention) and a control group (no intervention).

ELIGIBILITY:
Inclusion Criteria:

* Head and neck squamous cell carcinoma
* Indication for the protocol treatment of neoadjuvant chemotherapy followed by radiotherapy concomitant to chemotherapy.
* Oropharynges, larynx and hypopharynx advanced cancer (T3 or T4), classified as resectable;
* 18 years old or older;
* informed consent signed before any specific procedure

Exclusion Criteria:

* Previous head and neck surgery
* Previous radiotherapy or chemotherapy
* Previous history of neoplasia, excepted for in situ carcinoma of endometrial (uterine) cancer, skin basal cell or squamous cell carcinoma;
* Severe laryngeal aspiration during all consistencies swallowing evaluated thought videofluoroscopy
* Patients with cognitive deficit which could not comprehend the speech pathology intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-07; Primary Completion 2014-11 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Swallowing function | up to 6 months after concurrent phase.
  Self-reporting swallowing questionnaire, clinical swallowing examination and modified barium swallow (MBS), and the MD Anderson Dysphagia Inventory (MDADI).

CONTACTS AND LOCATIONS:
Overall Officials: André L Carvalho, PHD, Study Chair — Fundação Pio XII - Hospital de Câncer de Barretos; Luciano S Viana, PHD, Study Director — Fundação Pio XII - Hospital de Câncer de Barretos; Alexandre Jacinto, MD, Study Director — Fundação Pio XII - Hospital de Câncer de Barretos; Juliana Portas, MSC, Principal Investigator — Fundação Pio XII - Hospital de Câncer de Barretos
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil